CLINICAL TRIAL: NCT03138018
Title: The Potential Impact of Aging Stereotypes in the Assessment of Memory Deficits and Screening for Prodromal State of Alzheimer's Disease
Brief Title: Aging Stereotypes and Prodromal Alzheimer's Disease
Acronym: AGING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-45; IDRCB Number (Other: 2017-A00946-47)
Record Dates: First submitted 2017-04-10; First posted 2017-05-03 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard instruction (Active Comparator)
  Interventions: Diagnostic Test: Diagnosis of MCI versus No MCI (SCI or healthy patient)
- Reduced threat instruction (Experimental)
  Interventions: Diagnostic Test: Diagnosis of MCI versus No MCI (SCI or healthy patient)

INTERVENTIONS:
Diagnostic Test: Diagnosis of MCI versus No MCI (SCI or healthy patient) — Neuropsychological tests
Diagnostic Test: Diagnosis of MCI versus No MCI (SCI or healthy patient) — Neuroimaging biomarkers of neurodegeneration

SUMMARY:
Because of the lengthening of life expectancy, more and more people are concerned with the effects of aging on their mental faculties (e.g., memory decline) and with the possibility of getting Alzheimer's Disease (AD) or other forms of dementia. This increasing awareness of AD has already resulted in a growing demand for neuropsychological testing. AD's research also emphasizes the need for early screening to improve the prediction of the disease progression and the efficacy of any future therapy. Such a drive to screen for pre-dementia raises the challenging issue of frontline identification of individuals in the preclinical or early clinical stages of AD. Mild Cognitive Impairment (MCI) is typically considered to be the prodromal state of AD, and is therefore at the core of the drive for early screening. Moreover, Pre-MCI so called SCI (Subjective Cognitive Impairment) can precede AD for 15 years. However, many individuals diagnosed with MCI do not convert to AD, some remaining stable and others even reversing back to normal (with rates of reversion to normal varying from 4.5% to as high as 53%). This over-diagnosis bias, which has been largely overlooked, is at the core of the present project at the interface of human and life sciences. Here, we argue that an important source of overdiagnosis in the prodromal state of AD comes from negative aging stereotypes (e.g., the culturally shared beliefs that aging inescapably causes severe cognitive decline and diseases such as AD) that permeate neuropsychological screening. There is ample evidence in the laboratory that such stereotypes contribute to the differences observed in the healthy population between younger and older adults in explicit memory tasks. Additionally, three pilot (lab) studies specifically conducted for the present ANR project showed that the threat of being judged stereotypically undermines the controlled use of memory of healthy older adults and simultaneously intensifies their automatic response tendencies, resulting in impaired memory performance. The present proposal goes several steps further by examining for the first time whether aging stereotypes are powerful enough to implicitly permeate the clinical neuropsychological testing and thus inflate memory deficits in older adults judged "at risk" (based on either epidemiological criteria or memory complaints), resulting in false-positive detection of SCI and MCI. This provocative hypothesis will be tested while 1) using biomarkers of neurodegeneration to distinguish false-positives from true MCI, and 2) using biomarkers of stress to examine whether and how aging stereotypes can lead to acute physiological stress during neuropsychological testing. This innovative project has the potential to offer new recommendations to improve the diagnosis accuracy of prodromal state of AD, with positive consequences for older people's wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 50 years old
* Patients must report memory complaints
* Patients must show signs of MCI (amnestic single or multiple domain) on the following short cognitive tests

Exclusion Criteria:

* Probable Alzheimer's Disease according to NINCDS-ADRDA criteria (MA patients will be excluded from the study because false-positive errors only concern MCI status, not AD)
* Psychiatric disorders (schizophrenia, bipolar disorder)
* Cranial trauma
* Developmental pathologies
* Depression (score greater than or equal to 10 on GDS)
* Psychotropic medication if modified in the last 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological tests | 48 months
  Neuropsychological battery used for the diagnosis of Mild Cognitive Impairment (MCI, amnestic single or multiple domain)

SECONDARY OUTCOMES:
Neuroimaging biomarkers of neurodegeneration | 48 months
  Structural MRI (Hippocamp) and Florbetapir© PET (β-amyloid deposition)
Physiological stress | 48 months
  cortisol, dehydroepiandrosterone (DHEA) and its sulfated stable form (DHEAS) from the HPA axis, and Immunoglobulin A (IgA).
Self-report questionnaires | 48 months
  Vulnerability factors for stereotyping threat effects are assessed
Heart rate variability (thin elasticized heart rate transmitter belt), | 48 months
  Physiological stress
Skin conductance (wristwatch) | 48 months
  Physiological stress
Salivary biomarkers | 48 months
  cortisol, dehydroepiandrosterone (DHEA) and its sulfated stable form (DHEAS) from the HPA axis, and Immunoglobulin A (IgA).

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — ASSISTANCE PUBLIQUE HÔPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gauthier K, Morand A, Dutheil F, Alescio-Lautier B, Boucraut J, Clarys D, Eustache F, Girard N, Guedj E, Mazerolle M, Paccalin M, de la Sayette V, Zarea A, Huguet P, Michel BF, Desgranges B; AGING consortium; Regner I. Ageing stereotypes and prodromal Alzheimer's disease (AGING): study protocol for an ongoing randomised clinical study. BMJ Open. 2019 Oct 7;9(10):e032265. doi: 10.1136/bmjopen-2019-032265. PMID 31594904